CLINICAL TRIAL: NCT05342870
Title: A Sequential Allocation Study to Determine the ED50 of Dexmetedomidine as an Adjuvant to Lidocaine Intravenous Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Carine Zeeni, Assistant Professor, American University of Beirut Medical Center
Allocation: Not Applicable | Model: Sequential | Purpose: Treatment
Other Study IDs: ANES.CZ.01
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Bier Block; Dexmedetomidine; Tourniquet Pain; Carpal Tunnel; Tendon Release; Tendn Transfer
MeSH Terms: conditions — Median Neuropathy | interventions — Dexmedetomidine

STUDY DESIGN:
Masking Description: This is one arm non-randomized approach. Since it is a sequential approach of medication administration, the anesthesiologist and patients were blinded to whatever dose was given.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Following a sequential allocation scheme, the dexmedetomidine dose for each patient was determined by the Dixon up-and-down method. The dexmedetomidine dose for the first patient was 0.5 µg/kg. The dose was then adjusted in 0.1 µg/kg increments for the following patients depending on the success of the previous patient's block. If a patient experienced tourniquet pain prior to T0 + 50 minutes the next patient received a higher dose. If a patient did not experience pain at T0 + 50 minutes of tourniquet time the dose for the following patient was decreased. Identical syringes containing the solution mix were prepared by the principal investigator and handed to the blinded anesthesiologist in the room. Stopping rules were set at 6 independent crossovers in the same direction (no pain to pain or pain to no pain), with a minimum number of 20 patients

SUMMARY:
Intravenous Regional Anesthesia (IVRA) is an easy and reliable anesthetic technique for hand and forearm surgery. Its use is however limited by the presence of tourniquet pain during the surgery and the absence of postoperative analgesia. Many adjuvants to local anesthetics have been studied in order to overcome these shortcomings, including α2 adrenergic agonists. Clonidine has been shown to be efficacious when used with IVRA at a dose of 1µg/kg. Dexmetedomidine (DEX) is a recent more selective α2 adrenergic agonist that has been used successfully during IVRA at a dose of 0.5µg/kg. However when comparing potency ratios of Clonidine and DEX (8 to 1), the investigators hypothesize that a lower DEX dose would provide patients with adequate anesthesia.

We will determine the population average dose of DEX (ED50) that provides 50 minutes of tolerance to the tourniquet during a Lidocaine IVRA by a sequential Dixon up-down allocation study.

Eligible patients will be enrolled after obtaining informed consent. Patients will receive a standardized IVRA with Lidocaine and DEX adjuvant following a sequential allocation scheme. The first patient will receive a dose of 0.5 µg/kg of DEX. The dose will be then adjusted in 0.1 µg/kg increments for the following patients dependent on the success of the previous patients block. If a patient experiences tourniquet pain prior to 50 minutes after inflation of the distal tourniquet the next patient will receive a higher dose, if he does not experience pain prior to 50 minutes after inflation of the distal tourniquet the dose for the following patient will be decreased.

Recruitment will continue until 6 independent crossovers are observed with a minimum of 20 patients. The mean and the standard deviation of the ED50 of DEX will be calculated using the modified up-down method.

This study will help determine the ED50 of DEX used as an adjuvant in IVRA. Based on the potency ratios of Clonidine vs. DEX, the investigators hypothesize that the dose of DEX needed to achieve 50 minutes of pain free tourniquet time will be closer to 0.125 µg/kg rather than 0.5 µg/kg, a 75% reduction in the dose studied.

ELIGIBILITY:
Inclusion Criteria:

• Patients 18 to 70 years of age, ASA physical status I-II, undergoing unilateral hand or forearm surgery (that require 30 minutes or more) under IVRA.

Exclusion Criteria:

•Patients with Raynaud's disease, sickle cell anemia, heart block, allergy to any of the anesthetic drugs used, patients on α-adrenergic agonists, ASA III or IV, emergency surgery and pregnant patients., Weight greater than 100Kg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Median effective dose of dexmedetomidine | During the procedure
  The dexmedetomidine dose for the first patient was 0.5 µg/kg, the minimum tourniquet time chosen for our study was 50 minutes. The dose was then adjusted in 0.1 µg/kg increments for the following patients depending on the success of the previous patient's block. If a patient experienced tourniquet pain prior to T0 + 50 minutes the next patient received a higher dose. If a patient did not experience pain at T0 + 50 minutes of tourniquet time the dose for the following patient was decreased. Stopping rules were set at 6 independent crossovers in the same direction (no pain to pain or pain to no pain), with a minimum number of 20 patients. The mean and standard deviation of the ED50 of dexmedetomidine were calculated using the modified up-and-down method, which uses the average dexmedetomidine dose of all independent pairs of patients involved a crossover to calculate the ED50

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are not publicly available because the publicity policy is not yet generated by our institutional review board but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Karam C, Al Assadi S, Kanazi G, Zeeni C. A sequential allocation study to determine the ED50 of Dexmedetomidine as an adjuvant to lidocaine intravenous regional anesthesia. BMC Anesthesiol. 2022 May 27;22(1):165. doi: 10.1186/s12871-022-01702-9. PMID 35624418